CLINICAL TRIAL: NCT01606046
Title: Comparison of the Effects of Vapocoolant Spray and Topical Anesthetic Cream on Pain During Needle Electromyography: a Randomized Controlled Clinical Trial
Brief Title: Comparison of the Effects of Vapocoolant Spray and EMLA Cream on Pain During Needle Electromyography
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: The Catholic University of Korea (Other)
Responsible Party: Principal Investigator, Young Eun Moon, Clinical Professor, The Catholic University of Korea
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: momo0910
Record Dates: First submitted 2012-05-23; First posted 2012-05-25 (Estimated); Last update posted 2012-06-21 (Estimated); Status verified 2012-05

CONDITIONS: Electrodiagnosis
MeSH Terms: interventions — Lidocaine, Prilocaine Drug Combination

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (3):
- vapocoolant spray (Active Comparator)
  Interventions: Device: vapocoolant spray
- topical anesthetic agent (Active Comparator)
  Interventions: Drug: topical anesthetic cream
- Control (No Intervention): no interventions

INTERVENTIONS:
Device: vapocoolant spray — spray for 5 seconds from a distance of 30 cm just before the needle EMG
  Other Names: Ethyl chloride spray
  Arms: vapocoolant spray
Drug: topical anesthetic cream — application of EMLA cream on the needle electrode insertion site 60 minutes before the needle EMG
  Other Names: EMLA® (Eutectic Mixture of Local Anesthetics)
  Arms: topical anesthetic agent

SUMMARY:
The purpose of this study is to compare the effects of vapocoolant spray and topical lidocaine 2.5% + prilocaine 2.5% cream (EMLA) on reducing pain during needle electromyography.

DETAILED DESCRIPTION:
The study was conducted on patients with patients that underwent needle EMGs in the lower extremity between July and August 2011 at the university hospital. The patients were divided into a total of three groups by random assignment: a control group that did not receive pretreatment, a group that received ethyl chloride vapocoolant spray and a group that received topical anesthetic cream (EMLA cream®).The patients with spray group, they were sprayed with ethyl chloride vapocoolant spray for 5 seconds from a distance of 30 cm just before the needle EMG, and patients with EMLA cream, they received an application of topical anesthetic cream on the needle electrode insertion site 60 minutes before the needle EMG. The 37-mm monopolar needle electrode was vertically inserted into the medial head of the gastrocnemius muscle in all patients.

To assess the degree of pain for each group, patients were asked to indicate their level of pain on a 100 mm VAS (0, no pain; 100, worst intolerable pain) after the needle EMG in the gastrocnemius muscle.

In both experimental groups, a 5-point Likert scale was used to evaluate patient satisfaction with the pain reduction method used and their willingness to use the same analgesic method in another EMG.

ELIGIBILITY:
Inclusion Criteria:

* Patients who had a normal schedule of needle EMGs in the lower extremity.

Exclusion Criteria:

1. those who refused to participate in the experiment
2. those who were unable to understand a VAS and Likert scale
3. those with a history of allergic reaction to vapocoolant spray or lidocaine
4. those with a history of cold intolerance (Raynaud's syndrome, etc.)
5. those who took oral pain medications or used topical anesthetics within 24 hours of the experiment
6. those who exhibited abnormal lower extremity sensation during the physical examination or who showed pain on gastrocnemius

Ages: 19 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 99 (Actual)
Dates: Start 2011-07; Primary Completion 2011-07 (Actual); Study Completion 2011-08 (Actual)

PRIMARY OUTCOMES:
visual analogue scale, 5 point Likert scale | Immediately after the complete of needle electromyography

CONTACTS AND LOCATIONS:
Overall Officials: SangHyun Kim, Professor, Principal Investigator — Department of rehabilitation, Soon chun hyang university hospital Bucheon
Locations (1):
- Soonc chun hyang university hospital Bucheon, Bucheon-si, Gyeonngi-do, South Korea